CLINICAL TRIAL: NCT05792774
Title: Phrenic Afferences In Organic and Metabolic Illness: Central Sensitization - Fibromyalgia
Brief Title: Phrenic Nerve Infiltration in Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Angel Oliva Pascual-Vaca, Dr., University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PAINOMICS-fibromyalgia
Record Dates: First submitted 2023-03-19; First posted 2023-03-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: phrenic nerve; anesthesia, local; anesthetics; Pain; Bupivacaine
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phrenic nerve anesthetics infiltration (Experimental): The experimental intervention will consist of ultrasound-guided anesthetic blockade of the phrenic nerve at the laterocervical supraclavicular level with 1 ml of lidocaine without vasoconstrictor 2% to infiltrate the skin and 3ml of bupivacaine without vasoconstrictor 0.25% for neural blockade, making the local anesthetic surround the nerve between the anterior scalene muscle and the sternocleidomastoid muscle.
  Interventions: Drug: Bupivacain
- Physiological serum infiltration (Placebo Comparator): The placebo intervention will be similar in relation to 2% lidocaine without vasoconstrictor for the skin, but an ultrasound-guided puncture will be performed at the level of the subcutaneous cellular tissue by injecting 3 ml of physiological saline.
  Interventions: Other: Placebo (physiological saline serum infiltration)

INTERVENTIONS:
Drug: Bupivacain — The experimental intervention will consist of ultrasound-guided anesthetic blockade of the phrenic nerve at the laterocervical supraclavicular level with 1 ml of lidocaine without vasoconstrictor 2% to infiltrate the skin and 3ml of bupivacaine without vasoconstrictor 0.25% for neural blockade, making the local anesthetic surround the nerve between the anterior scalene muscle and the sternocleidomastoid muscle.
  Other Names: Bupivacaine B. Braun 2.5 mg/ml
  Arms: Phrenic nerve anesthetics infiltration
Other: Placebo (physiological saline serum infiltration) — The placebo intervention will be similar in relation to 2% lidocaine without vasoconstrictor for the skin, but an ultrasound-guided puncture will be performed at the level of the subcutaneous cellular tissue by injecting 3 ml of physiological saline.
  Arms: Physiological serum infiltration

SUMMARY:
It is known that nociceptive afferences in visceral pain and visceral disorders increase sensitization in subjects suffering from fibromyalgia. These patients use to present visceral comorbidities. Those comorbidities include that of peridiaphragmatic organs, which are supplied by the phrenic nerve among other innervations. It is known that peridiaphragmatic organs trigger referred pain in the neck area, via the phrenic nerves. So, the phrenic nociceptive afferences can be contributing to enhance the state of sensitization in fibromyalgia. This study aims to analyze the ability of phrenic nerve infiltration to diminish sensitization in subjects suffering fibromyalgia, by means of a randomized controlled trial.

DETAILED DESCRIPTION:
Fibromyalgia is a major problem due to issues such as the impact on quality of life and the associated health and social costs. It is characterized by a generalized state of sensitization, with a high level of perceived pain, among other features. Peripheral pain sources potentially exacerbate the central sensitization and its symptoms of chronic diffuse musculoskeletal pain and hyperalgesia. It has been shown that visceral pain enhances the level of central sensitization typical of the syndrome. So, it has been claimed that systematic assessment and treatment of visceral pain comorbidities should be a part of the management strategy in fibromyalgia.

Patients with fibromyalgia present visceral comorbidities. Those comorbidities include that of peridiaphragmatic organs, which are supplied by the phrenic nerve among other innervations. It is known that peridiaphragmatic organs trigger referred pain in the neck area, via the phrenic nerves. So, the phrenic nociceptive afferences can be contributing to enhance the state of sensitization in fibromyalgia. This study aims to analyze the ability of phrenic nerve infiltration to diminish sensitization in subjects suffering fibromyalgia.

For this purpose, the investigators intend to perform a randomized clinical trial, assessing the effects on pain threshold to pressure, visual analogue scale, range of motion and fibromyalgia specific questionnaires. There will be only one intervention session. The experimental group will receive an ultrasound-guided anaesthetic infiltration of the phrenic nerve, while the control group will receive a placebo infiltration. A one-week follow-up, with intermediate measurements, will be carried out to assess the evolution of sensitization and symptomatology.

The results of this study will make it possible to establish the role of phrenic afferences in fibromyalgia sensitization, thus making it possible to specify a specific therapeutic target (phrenic nerve) as well as the importance of visceral treatment in subjects with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Over 18 and under 64 years old
* Diagnosis of Fibromyalgia
* Any peridiaphragmatic visceral disorder diagnosed by the respective specialist.
* That the subject agrees to participate in the project by signing the informed consent.

Exclusion Criteria:

* Other rheumatic diseases.
* Degenerative neurological disease.
* Major psychiatric disorder
* Cognitive deterioration
* Non-cooperative subject
* Any medical condition affecting sensory evaluation
* Contraindication to infiltration of the phrenic nerve.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Algometry | Pre-intervention. Post-intervention: 1 hour, 3 days and 7 days
  Pressure pain threshold in the specific 18 tender points in fibromyalgia. PPT levels defined as the minimum necessary pressure to evoke pain will be evaluated using a handheld electronic pressure algometer. Change from baseline in algometry.

SECONDARY OUTCOMES:
Patient Global Impression of Improvement | Pre-intervention. Post-intervention: 1 hour, 3 hours, 6 hours, 9 hours, 24 hours, 2 days, 3 days and 7 days
  Patient Global Impression of Improvement (PGI-Improvement) scale, ranging from 1 (very much better) to 7 (very much worse). It will be assessed verbally.
Numeric Pain Rating Scale | Pre-intervention. Post-intervention: 1 hour, 3 hours, 6 hours, 9 hours, 24 hours, 2 days, 3 days and 7 days
  Perceived pain. Self-perceived pain intensity will be evaluated by a 0 to 10 Numeric Pain Rating Scale (NPRS), where 0 denotes no pain and 10 denotes the maximum possible pain.
Fibromyalgia Survey Questionnaire | Pre-intervention. Post-intervention: 7 days.
  Fibromyalgia Survey Questionnaire (Questionnaire) (parts I and III). The Fibromyalgia Survey Questionnaire will be used in the Spanish version. This questionnaire assesses the severity of fibromyalgia symptoms. The first part of this questionnaire is constituted by 3 questions related to the last week, and they have to be answered by likert scales of 3 points. Higher scores indicate higher disability. The third part of this questionnaire is constituted by a qualitative localization of pain in the last week. A higher number of body regions suffering pain constitute a worse outcome. Parts II and IV of the questionnaire will not be considered as an outcome measure since they evaluate periods of 6 months and 3 months respectively, and our post-intervention measurement will be performed just 7 days after intervention, so these parts of the questionnaire have no interest as outcome measures.
Revised Fibromyalgia Impact Questionnaire | Pre-intervention. Post-intervention: 7 days.
  Revised Fibromyalgia Impact Questionnaire (Questionnaire). This questionnaire evaluates the difficulty to develop certain daily-life activities. It will be used in the Spanish version. This questionnaire assesses the severity of fibromyalgia symptoms. Scores range from 0-100 with higher scores indicating higher disability.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Oliva Pascual-Vaca, Dr, Principal Investigator — University of Seville
Locations (4):
- Spain (4):
  - Nacho Navarro Fisioterapia, Dos Hermanas, Seville
  - Asociación de Fibromialgia de Lebrija, Lebrija, Seville
  - Asociación de Fibromialgia de Sevilla, Seville, Seville
  - Hospitales Universitarios Virgen del Rocío y Macarena, Seville

IPD SHARING:
Plan to Share IPD: No